CLINICAL TRIAL: NCT01010880
Title: A Phase I/IIA, Non-Randomized, Open Label, Single Dose, Dose-Escalation, Safety Study of BKT140, a CXCR4 Antagonist in Patients With Multiple Myeloma
Brief Title: Safety Study of a Chemokine Receptor (CXCR4) Antagonist in Multiple Myeloma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biokine Therapeutics Ltd (Industry)
Responsible Party: Dr Orly Eizenberg, Biokine Therapeutics Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BKTSC001
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; CXCR4; Stem Cells; Mobilization; Transplantation; Chemotherapy
MeSH Terms: conditions — Multiple Myeloma | interventions — BKT140

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: BKT140 — BKT-140 drug substance is a highly selective CXCR4 antagonist. BKT140 will be injected S.C once at dose of 0.03, 0.1, 0.3, 0.9 mg/kg

SUMMARY:
BKT-140 drug substance is a highly selective chemokine receptor (CXCR4) antagonist, which is developed by Biokine as a novel therapy for Multiple Myeloma (MM, a type of blood cancer). The unique combination of activities of BKT140, i.e., the induction of the exit of blood cells such as stem cells and mature cells from the bone marrow to the peripheral blood, coupled with specific induction of MM cell death by BKT-140, represents a novel therapeutic strategy against MM.

DETAILED DESCRIPTION:
The chemokine CXCL12 (also called SDF-1 - stromal-derived-factor-1) and its receptor, CXCR4 ((CXC Chemokine Receptor 4), a molecule endowed with potent chemotactic activity for hematopoietic cells, together play a pivotal role in the trafficking of hematopoietic stem cells to the bone marrow 10,11. The CXCL12/CXCR4 axis is also critically involved in the retention of hematopoietic cells within the BM microenvironment. Following chemotherapy and irradiation, the CXCL12/CXCR4 axis delays the recovery of the BM progenitor cells and the exit of mature cells such as neutrophils and monocytes to the periphery. Consequently, disruption of the CXCL12/CXCR4 interaction results in mobilization of hematopoietic cells including stem cells and a faster recovery of the treated BM.

BKT140 (4F-benzoyl-TN14003) is a highly selective and unique CXCR4 antagonist. Pre-clinical studies showed that BKT140 binds CXCR4 with high affinity (1nM) 13. Biokine has demonstrated the ability of the CXCR4 antagonist, BKT140, to mobilize various WBC such as neutrophils and monocytes as well as progenitor and stem cells, from the BM. The ability of BKT140 to stimulate the mobilization of these cells is superior to that of AMD3100, a CXCR4 antagonist that is in clinical development for mobilization of stem cells in MM and lymphoma patients, both qualitatively and quantitatively. BKT140 synergizes much more efficiently with G-CSF when compared to AMD3100. Moreover, Biokine has shown that BKT140, in synergism with G-CSF (NEUPOGEN®), is much more efficient in increasing the numbers of neutrophils and activated monocytes in the blood, by several folds as compared to G-CSF alone. BKT140 also shortens the neutropenic period due to an early release of neutrophils and monocytes from the BM. More importantly, BKT140, in synergism with G-CSF, reduces the anemic period caused by chemotherapy, due to a RBC production, which does not occur when G-CSF is given as a sole treatment. More importantly, BKT140, but not G-CSF or AMD3100, is also capable of shortening the period of cytopenia by boosting both the recovery of all hematopoietic cells in the BM and their exit to the periphery, and therefore shortening the period of cytopenia following chemotherapy or irradiation and BM transplantation. Importantly, Biokine has shown that upon interaction with CXCR4, BKT140, but not AMD3100, selectively, specifically and rapidly stimulates human leukemia and myeloma cell death in vitro and in vivo. Furthermore, BKT140 synergizes with other chemotherapeutic agents such as rapamycine to induce MM cell death.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 to 65 years old inclusive
* MM patients with clinically significant disease that achieved at least Partial Response (PR) after induction chemotherapy
* Patients eligible for HDC with PBSC support.
* Patients who require stem cell collection with CTX and G-CSF priming.
* Normal LV functions (EF over 50%, DLCO over 50%)
* Karnofsky score > 60%,
* Patients must have normal renal and liver functions as defined below:

  * Total bilirubin ≤2.0 x institutional upper limit of normal (ULN), unless the patient has a known diagnosis of Gilbert's disease.
  * Aspartate transaminase (AST, SGOT) or alanine transaminase (ALT, SGPT) ≤3 x institutional ULN.
  * Serum creatinine ≤1.5 g/dL or calculated estimated creatinine clearance ≥40 mL/min
* Polymorphonuclear neutrophil (PMN) count > 1,500
* PLT >100,000
* Hemoglobin > 9gr%
* Women of child-bearing potential must have a negative serum or urine pregnancy test at enrollment.
* If female, the patient is post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (e.g., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide or abstinence) from the enrollment visit through 30 days after the administration of the study drug.
* If male, the patient agrees to use an acceptable barrier method of contraception from the time of enrollment through 30 days after the administration of the study drug.
* Prior to enrollment, the patient is capable of understanding the protocol and able to sign a written informed consent.

Exclusion Criteria:

* Patients who have not achieved at least Partial Response (PR) following induction chemotherapy.
* No pervious G-CSF therapy.
* Creatinine clearance <40 mL /min.
* Body temperature above 385 C on day 10.
* Patients with blood pressure <105/60
* Any of the following in the last 3 months prior to enrollment: Unstable Angina, Acute Myocardial Infarction (MI), Congestive Heart Failure, CVA, uncontrolled blood pressure
* Pregnant or breast-feeding women.
* Any medical condition which in the opinion of the Investigator places the patient at an unacceptably high risk for toxicities.
* Treatment with any investigational agents in the last 21 days before study entry.
* Any condition or circumstance which, in the opinion of the Investigator, would significantly interfere with the patient's protocol compliance and put the patient at increased risk.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
White blood cell (WBC) count | 24 hour

SECONDARY OUTCOMES:
CD34+ cells | 24 hour

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (2):
- Israel (2):
  - Department of Hematology and Bone Marrow Transplantation,Rambam Medical Center, Haifa
  - Chaim Sheba Medical Center,Tel-Hashomer, Ramat Gan

REFERENCES:
- [Background] Abraham M, Biyder K, Begin M, Wald H, Weiss ID, Galun E, Nagler A, Peled A. Enhanced unique pattern of hematopoietic cell mobilization induced by the CXCR4 antagonist 4F-benzoyl-TN14003. Stem Cells. 2007 Sep;25(9):2158-66. doi: 10.1634/stemcells.2007-0161. Epub 2007 May 24. PMID 17525235